CLINICAL TRIAL: NCT06596213
Title: Overcoming Inequalities in Health to Eliminate Hepatitis - Real-World Evidence from a Territory-Wide Cohort
Brief Title: Hepatitis Inequalities Study
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Other Study IDs: CRE2024.361
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Chronic Hepatitis B; HEPATITIS C VIRUS CHRONIC INFECTION
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Health inequality in liver diseases including age, gender, ethnicity and socioeconomic status has been increasingly recognised and potentially hinder hepatitis elimination. Health inequality has significant impact to evaluate the impact diagnostic and treatment uptake rates of chronic viral hepatitis on risk of hepatocellular carcinoma (HCC), hepatic event and liver-related death in patients with chronic hepatitis B and/or C. To overcome the limitation of small prospective cohort study of limited recruitment period, retrieving information from the Clinical Data Analysis and Reporting System (CDARS) from Hospital Authority (HA) will be one of the best way to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have any of these viral markers (HBeAg / HBsAg / HBV DNA / HCV RNA) and/or any of the following diagnosis codes (ICD-9 070-070.9; 348.3, 349.82, 456, 456.2, 456.8, 567.2, 567.8, 570, 571.2, 571.5, 571.6, 572.2, 572.3, 572.4, 789.5) checked or coded in any public hospitals or clinics from 1 January 2000 to 31 March 2024.

Exclusion Criteria:

* Patients with missing age, gender, ethnicity and socioeconomic status
* (Subgroup analysis for ethnicity and socioeconomic status) Patients with missing ethnicity and socioeconomic status
* Serious medical illnesses or malignancy with life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From the Clinical Data Analysis and Reporting System (CDARS) from Hospital Authority
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety | From 1 January 2000 to 31 March 2024
  Time from diagnosis of hepatitis to treatment.

SECONDARY OUTCOMES:
Safety | From 1 January 2000 to 31 March 2024
  The composite endpoints of recurrence of hepatic events (e.g. HCC hepatic coma, portal hypertension, variceal bleeding, hepatorenal syndrome).

REFERENCES:
- [Background] El-Serag HB. Epidemiology of viral hepatitis and hepatocellular carcinoma. Gastroenterology. 2012 May;142(6):1264-1273.e1. doi: 10.1053/j.gastro.2011.12.061. PMID 22537432
- See also: Hepatitis B — https://www.chp.gov.hk/en/healthtopics/content/24/27.html